CLINICAL TRIAL: NCT04280666
Title: An Exploratory Study of Next-generation Sequencing in Colorectal Cancer Somatic Cells to Guide Screening for Genetic Susceptibility Gene Mutations.
Brief Title: Next-generation Sequencing of Colorectal Cancer Somatic Cells to Guide Genetic Susceptibility Gene Mutations Screening.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Fangqi Liu, Dr., Fudan University
Other Study IDs: FDCRC49-LFQ
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Hereditary Colorectal Cancer
Keywords: Colorectal Cancer; Next-generation sequencing; Genetic Susceptibility
MeSH Terms: conditions — Colorectal Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and formalin-fixed tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, single-center, clinical study.This study is to evaluate the feasibility of genetic susceptibility screening based on the detection of tumor tissue mutations by a NGS panel.

DETAILED DESCRIPTION:
In this study, gene mutation profiling was performed on primary tissue samples from colorectal cancer patients who met relevant clinical screening criteria, unearthing suspected germline pathogenic mutations. At the same time, germline mutation detection was performed on peripheral blood leukocytes of patients, and the consistency between suspected germline mutations in tumor somatic mutation detection and control leukocytes was compared. Establishing the feasibility of tumor somatic mutation-based detection to guide genetic susceptibility screening.Pedigree verification will be carried out for blood relatives of patients with germline mutations which have been identified for colorectal cancer.Through the tumor somatic and germline gene mutation profiles of Chinese hereditary colorectal cancer patients, it reveals the molecular characteristics of hereditary colorectal cancer in Asian populations and provides molecular-level evidence for possible subsequent clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* A biopsy proven histological diagnosis of colorectal carcinoma.
* ≥ 18 years of age on the day of signing informed consent.
* Patients must meet the relevant clinical screening standards, such as the Amsterdam Standard (I / II),etc.
* Patients need to provide tumor tissue samples and matched peripheral blood (leukocyte) samples.

Exclusion Criteria:

* History of other malignant tumors(except for cervical carcinoma in situ, basal or squamous cell skin cancer which has been fully treated).
* There is no detailed histopathological report to judge the nature of the lesions.
* Any social or psychological problems, etc., which are judged by the researcher to be unsuitable for the study.
* For various reasons, the baseline samples (tumor tissue samples, peripheral blood samples) were incomplete.
* Patients who are unwilling or unable to follow the research program for long-term and regular follow-up in current medical institutions.
* Failure to complete the follow-up within 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients who meet the relevant clinical screening standards (such as Amsterdam standard (I / II), Bethesda standard (Revised Version) and China expert consensus on clinical diagnosis, treatment and family management of hereditary colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity, specificity, positive predictive value, and negative predictive value | 1.5 years
  Assessing the sensitivity, specificity, positive predictive value, and negative predictive value of genetic susceptibility gene mutations screening based on a targeted Next-generation sequencing panel.

SECONDARY OUTCOMES:
pedigree verification of candidate patients | 3.5 years
  Screening for leukocyte mutations in blood relatives of the hereditary colorectal cancer patients with germline mutations.Preliminary analysis of the distribution, clinical characteristics, molecular typing and prognosis of Chinese hereditary colorectal cancer patients and their families.
Characteristics of the gene map and the correlations with clinical characteristics | 3.5 years
  Gene map characteristics of tissue samples from colorectal cancer patients who meet the relevant clinical screening criteria and their correlations with clinical characteristics (age, gender, family history, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai, China